CLINICAL TRIAL: NCT03466736
Title: Enriching Clinical Trials Requiring Amyloid Positivity With Practice Effects
Acronym: APPE
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kevin Duff, Professor of Neurology, University of Utah
Other Study IDs: R01AG055428 (NIH)
Record Dates: First submitted 2018-03-07; First posted 2018-03-15 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: practice effects; amyloid imaging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cognitively intact older adults: Each subject will receive an amyloid PET scan with [18F]flutemetamol
  Interventions: Diagnostic Test: [18F]flutemetamol PET scan
- Mild Cognitive Impairment: Each subject will receive an amyloid PET scan with [18F]flutemetamol
  Interventions: Diagnostic Test: [18F]flutemetamol PET scan
- Alzheimer's disease: Each subject will receive an amyloid PET scan with [18F]flutemetamol
  Interventions: Diagnostic Test: [18F]flutemetamol PET scan

INTERVENTIONS:
Diagnostic Test: [18F]flutemetamol PET scan — Each subject will receive an amyloid PET scan with [18F]flutemetamol

SUMMARY:
The primary objective of this study is to demonstrate that individuals with low short-term practice effects (STPE) on cognitive testing are more likely to be identified as "positive" on amyloid imaging than individuals with high STPE. STPE may also inform us about other AD-related biomarkers, including hippocampal volumes, functional connectivity, and APOE status. By realizing the aims of this pragmatic study, we hope to be able to offer more economical and efficient screening of potential participants for clinical trials, which would reduce participant burden and financial costs.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Identified as intact, Mild Cognitive Impairment, or Alzheimer's disease
* Able to complete study procedures
* All participants must have a collateral source (e.g. spouse, adult child, caregiver, close friend) available to briefly comment on the cognitive abilities and daily functioning of the participant. If the participant is diagnosed with probable AD dementia, a legally authorized representative (e.g. spouse, adult child) must be available to provide informed consent for the participant.

Exclusion Criteria:

* History of major stroke, head injury with loss of consciousness of >30 minutes, or other neurological/systemic illness that may affect cognition
* Current or past major psychiatric illness (e.g., schizophrenia, bipolar affective disorder)
* History of substance abuse
* Current use of antipsychotics or anticonvulsant medications
* Known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals.
* Need for monitored sedation or anesthesia during PET or MRI scanning.
* Claustrophobia to a degree that the individual cannot undergo PET or MRI imaging
* History of metal injury which precludes the individual from undergoing MRI imaging
* Evidence of stroke or mass lesion on a CT or MRI scan
* History of radiation therapy to the brain
* History of significant major medical illnesses, such as cancer or AIDS.
* Inadequate vision, hearing, and manual dexterity to participate in the cognitive assessments.
* 15-item Geriatric Depression Scale score of >5
* Clinical Dementia Rating score of >1
* Mini Mental State Examination score of <20

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults who are either cognitively intact, have Mild Cognitive Impairment, or have Alzheimer's disease
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
short-term practice effects | baseline and one week
  Amount of improvement when cognitive tests are repeated twice within one week

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duff K, Dixon AM, Embree L, Hoffman JM. Change on the Repeatable Battery for the Assessment of Neuropsychological Status and its relationship to brain amyloid. J Clin Exp Neuropsychol. 2023 Mar;45(2):105-117. doi: 10.1080/13803395.2023.2216920. Epub 2023 May 24. PMID 37224404
- [Derived] Duff K. Revisiting reliable change with Iverson (2001). Clin Neuropsychol. 2024 Feb;38(2):412-428. doi: 10.1080/13854046.2023.2202333. Epub 2023 Apr 20. PMID 37081822
- [Derived] Duff K, Wan L, Embree L, Hoffman JM. Change in the Quick Dementia Rating System Across Time in Older Adults with and without Cognitive Impairment. J Alzheimers Dis. 2023;93(2):449-457. doi: 10.3233/JAD-221252. PMID 37038819
- [Derived] Duff K, Wan L, Levine DA, Giordani B, Fowler NR, Fagerlin A, King JB, Hoffman JM. The Quick Dementia Rating System and Its Relationship to Biomarkers of Alzheimer's Disease and Neuropsychological Performance. Dement Geriatr Cogn Disord. 2022;51(3):214-220. doi: 10.1159/000524548. Epub 2022 Apr 27. PMID 35477163
- [Derived] Duff K, Suhrie KR, Dalley BCA, Porter SM, Dixon AM. Recognition subtests for the Repeatable Battery for the Assessment of Neuropsychological Status: Preliminary data in cognitively intact older adults, amnestic Mild Cognitive Impairment, and Alzheimer's disease. Clin Neuropsychol. 2021 Nov;35(8):1415-1425. doi: 10.1080/13854046.2020.1812724. Epub 2020 Sep 3. PMID 32883179